CLINICAL TRIAL: NCT05169034
Title: Feasibility of Predicting Blood Glucose Values by Measuring in the Interstitial Fluid of the Skin on the Wrist With the Non-invasive Medical Device D-Base
Brief Title: Feasibility Study of Blood Glucose Monitoring With the Non-invasive Medical Device D-Base
Status: Terminated | Type: Observational
Why Stopped: Goals as defined in the study protocol were not met after the first study period. Study with improved device will follow.
Sponsor: Diamontech AG (Industry)
Collaborators: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Responsible Party: Sponsor
Other Study IDs: IfDT-2012-DE
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to evaluate the feasibility of monitoring the blood glucose values by measuring the glucose in the interstitial fluid of the skin on the wrist of subjects with diabetes mellitus type 1 and 2.

DETAILED DESCRIPTION:
The investigation is designed as an open, monocentric, non-randomized, single-arm, explorative study in adult subjects with type 1 or 2 diabetes mellitus (any therapy form).

The clinical investigation will be performed in an outpatient setting on up to two study days with up to 100 subjects. A nearly equal number of subjects with diabetes type 1 and 2 shall participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 or type 2 diabetes
* HbA1c <10%
* An understanding of and willingness to follow the protocol
* Signed informed consent

Exclusion Criteria:

* Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment
* Hypoglycemia unawareness
* Have extensive skin changes/diseases at the proposed measurement site (wrist) that could interfere with the accuracy of glucose measurements.
* Female subjects: pregnancy, lactation period, lack of a negative pregnancy test (except in case of menopause, sterilization or hysterectomy)
* Serious acute or chronic disease besides diabetes mellitus or an anamnesis which might, in the opinion of the investigator, pose a risk to the subject, e.g. seizure disorder, adrenal disorder, dialysis for renal failure, cystic fibrosis, active infection
* Severe diabetes related complications (i.e. severe macro angiopathy, severe micro angiopathy, severe neuro-, retino- or nephropathy) when unstable (defined by event or increasing symptoms in the last 6 months) or with insufficient therapy
* Any incapacity or general condition that, in the opinion of the investigator, prevents adequate compliance with the study procedures, e.g. mental or visual incapacity, tremor, language barriers, alcohol or drug misuse
* Not able to understand, write or read German
* Dependency from the sponsor or the clinical investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 adults with type 1 or type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
System Performance | 1 week per subject
  Accuracy of glucose values determined with the device in comparison with values from a standard glucometer

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Baden-Wurttemberg, Germany